CLINICAL TRIAL: NCT01399970
Title: Use of Mobile Teledermatology in the Care of Acne Patients - A Randomized Controlled Trial
Brief Title: Use of Mobile Teledermatology in the Care of Acne Patients
Acronym: Teleacne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: National Bank of Austria (Other Government)
Responsible Party: Principal Investigator, Rainer Hofmann-Wellenhof, MD, Prof. Dr., Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 02
Record Dates: First submitted 2011-04-27; First posted 2011-07-22 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Acne
Keywords: Mobile Teledermatology; Telemedicine; Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Pemetrexed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Outpatient Consultation Arm (OCA) (Other): Conventional in Office Care
  Interventions: Other: Outpatient Consultation Arm (OCA)
- Mobile Teleconsultation Arm (MTA) (Experimental): Mobile Teledermatology Care
  Interventions: Other: Mobile Teleconsultation Arm (MTA)

INTERVENTIONS:
Other: Mobile Teleconsultation Arm (MTA) — In addition to a face-to-face visit at baseline, patients will conduct "mobile visits" at home every two weeks. The general practitioner of choice will perform examinations, such as laboratory or occasionally pregnancy tests every 4 weeks according to the treatment guidelines.
  Other Names: MTA; Health Care Service Modality
  Arms: Mobile Teleconsultation Arm (MTA)
Other: Outpatient Consultation Arm (OCA) — Patients will receive routine outpatient care at the clinic according to the treatment guidelines, and will be scheduled for outpatient visits every 4 weeks.
  Other Names: OCA; Health Care Service Modality
  Arms: Outpatient Consultation Arm (OCA)

SUMMARY:
The purpose of the present study is to determine whether a mobile teledermatology care model can achieve better clinical outcomes as compared to conventional, outpatient care for the management of severe acne treated with isotretinoin.

The superiority of mobile care in comparison to conventional, outpatient care will be investigated regarding

1. effectiveness: Global evaluation Acne (GEA) score -response at week 24
2. safety: drop out rates and medication side effects
3. overall patient satisfaction with acne care and therapy
4. overall physician satisfaction with mobile acne care

ELIGIBILITY:
Inclusion Criteria:

Female or male, aged 12 to 30 years

* with facial acne
* requiring systemic isotretinoin treatment (GEA-Score: 3-5)
* with basic handy skills
* with a signed consent form

Exclusion Criteria:

* Pregnancy or lactation period
* Withdrawal of informed consent
* Non-compliance, failure to comply with protocol requirements

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 69 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Global evaluation Acne score (GEA) | week 24
  Change from Baseline in the median GEA score at week 24

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Hofmann-Wellenhof, MD, Study Director — Department of Dermatology, Medical University of Graz
Locations (1):
- Department of Dermatology, Medical University of Graz, Graz, Graz, Austria